CLINICAL TRIAL: NCT05201534
Title: Interventions in Math Learning Disabilities: Cognitive and Neural Correlates
Brief Title: Interventions in Mathematics and Cognitive Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Vinod Menon, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62479; 2R01HD059205-11A1 (NIH); SPO #42749 (Other Grant/Funding Number: Stanford Sponsored Projects Number)
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Math Learning Disability; Child Development; Developmental Disability; Learning Disabilities; Learning Disabled; Learning Curve; Mathematics Disorder; Dyscalculia; Dyscalculia, Primary; Dyscalculia, Acquired; Specific Learning Disorder, With Impairment in Mathematics; Individuality; Behavior, Child; Behavior and Behavior Mechanisms; Behavior; Decision Making; Neuronal Plasticity; Cognition; Cognition Disorder; Cognitive Dysfunction; Cognitive Change; Cognitive Impairment, Mild; Cognitive Developmental Delay; Cognitive Orientation; Cognitive Delay, Mild; Cognitive Deficits, Mild; Cognitive Abnormality; Neuroscience
Keywords: Numerical skills in children; Low math abilities; Mathematical Learning Disabilities; Mathematical Concepts; Mathematics; Transfer, Psychology; Generalization, Psychology; Early Intervention, Educational; Neural Pathways; Neural Networks, Computer
MeSH Terms: conditions — Dyscalculia; Developmental Disabilities; Learning Disabilities; Specific Learning Disorder; Child Behavior; Behavior; Cognition Disorders; Cognitive Dysfunction; Orientation, Spatial; Lymphoma, Follicular | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrative Symbolic Non-Symbolic (iSNS) Training (Experimental): Integrative symbolic non-symbolic (iSNS) training: Over a period of 6 weeks, participants will complete activities that progressively strengthen the mapping of symbolic numerical representations to non-symbolic numerical quantities and enhance fluency in symbolic numerical skills.
  Interventions: Other: Interventions in Mathematics and Cognitive Skills - Experimental
- Active Comparator: Active Control Intervention (Working Memory Training) (Active Comparator): Active control intervention: Over a period of 6 weeks, participants will complete activities that enhance short-term storage and maintenance of visuospatial or verbal information.
  Interventions: Other: Interventions in Mathematics and Cognitive Skills - Active Comparator

INTERVENTIONS:
Other: Interventions in Mathematics and Cognitive Skills - Experimental — After study participants have completed screenings to meet our inclusion criteria, participants will take part in the pre-training MRI brain scan (if eligible) and behavioral assessments and will then be assigned to the intervention for 6 weeks.
  During this training, participants will spend three days each week completing a set of problems at their home on a tablet that we provide them. Participants will receive one-to-one training with a member of our research team once a week.
  Following the completion of the 6-week training program, participants will be asked to complete a second MRI brain imaging session (for those who completed pre-training MRI) and post-measure appointments in order to assess immediate effects of the training program. Participants will also be invited to return for follow-up testing after six months in order to assess the long- lasting effects of the training program.
  Arms: Integrative Symbolic Non-Symbolic (iSNS) Training
Other: Interventions in Mathematics and Cognitive Skills - Active Comparator — After study participants have completed screenings to meet our inclusion criteria, participants will take part in the pre-training MRI brain scan (if eligible) and behavioral assessments and will then be assigned to the intervention for 6 weeks.
  During this training, participants will spend three days each week completing a set of problems at their home on a tablet that we provide them. Participants will receive one-to-one training with a member of our research team once a week.
  Following the completion of the 6-week training program, participants will be asked to complete a second MRI brain imaging session (for those who completed pre-training MRI) and post-measure appointments in order to assess immediate effects of the training program. Participants will also be invited to return for follow-up testing after six months in order to assess the long- lasting effects of the training program.
  Arms: Active Comparator: Active Control Intervention (Working Memory Training)

SUMMARY:
The purpose of this study is to investigate neurocognitive mechanisms underlying response to intervention aimed at enhancing, and remediating weaknesses in, numerical skills in children, including those with mathematical learning disabilities (MLD).

DETAILED DESCRIPTION:
The purpose of this study is to investigate neurocognitive mechanisms underlying response to intervention aimed at enhancing, and remediating weaknesses in, numerical skills in children, including those with mathematical learning disabilities (MLD).

To achieve this goal, investigators will use a theoretically-motivated integrated symbolic/non-symbolic (iSNS) intervention with a randomized controlled design to enhance cross-format mapping between symbolic and nonsymbolic representations of quantities. The investigators will develop innovative computational models to investigate individual differences in latent cognitive processes and brain plasticity that contribute to learning, long-term retention, and transfer in children.

The investigators will assess performance in several areas and investigate cognitive and neural mechanisms that support numerical skill acquisition in children with differing levels of math learning abilities.

ELIGIBILITY:
Inclusion Criteria:

1. Elementary school aged children starting from first grade (6-12 years old)
2. IQ: Participants with a Full Scale IQ > 70 on the Wechsler Abbreviated Scle of Intelligence (WASI-II).
3. Identification of Mathematical Learning Disabilities: Scores below the 35th percentile percentile on symbolic number processing test in Numeracy Screener and two or more Wechsler Individual Achievement Test (WIAT-IV) math subtests
4. Identification of typically developing children: Scores at or above the 35th percentile percentile on symbolic number processing test in Numeracy Screener and all WIAT-IV math subtests
5. Normal or corrected-to-normal vision and no hearing impairments
6. Inclusion in MRI scan session: Right-handed

Exclusion Criteria:

1. History of neurological or psychiatric disorder (i.e., schizophrenia, psychosis, depression, or attention deficit hyperactivity disorder.)
2. History of trauma involving head injury
3. Consistent psychiatric medications
4. Exclusion from MRI scan session: No major contraindication for magnetic resonance imaging (MRI) - braces, metal implants, pacemakers, vascular stents, metallic ear tubes, consistent exposure to metal, claustrophobia)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in symbolic number comparison task performance (reaction time) | Baseline and post-intervention (after 6 weeks)
  Performance will be measured by children's reaction time (milliseconds) on symbolic number comparison task
Change from baseline in symbolic number comparison task performance (accuracy) | Baseline and post-intervention (after 6 weeks)
  Performance will be measured by children's accuracy (% trials correct) on symbolic number comparison task
Change from baseline in non-symbolic number comparison task performance (reaction time) | Baseline and post-intervention (after 6 weeks)
  Performance will be measured by children's reaction time (milliseconds) on non-symbolic number comparison task
Change from baseline in non-symbolic number comparison task performance (accuracy) | Baseline and post-intervention (after 6 weeks)
  Performance will be measured by children's accuracy (% trials correct) on non-symbolic number comparison task
Change from baseline in latent cognitive measures of symbolic number comparison task performance (drift rate) | Baseline and post-intervention (after 6 weeks)
  Latent cognitive processing will be measured by drift rate from children's symbolic number comparison task performance
Change from baseline in latent cognitive measures of symbolic number comparison task performance (post-error adjustment) | Baseline and post-intervention (after 6 weeks)
  Latent cognitive processing will be measured by post-error adjustment from children's symbolic number comparison task performance
Change from baseline in latent cognitive measures of non-symbolic number comparison task performance (drift rate) | Baseline and post-intervention (after 6 weeks)
  Latent cognitive processing will be measured by drift rate from children's non-symbolic number comparison task performance
Change from baseline in latent cognitive measures of non-symbolic number comparison task performance (post-error adjustment) | Baseline and post-intervention (after 6 weeks)
  Latent cognitive processing will be measured by post-error adjustment from children's non-symbolic number comparison task performance
Change from baseline in brain activation during symbolic number comparison task performance | Baseline and post-intervention (after 6 weeks)
  Neural activity will be measured during functional magnetic resonance imaging (fMRI) symbolic number comparison task. Data will consist of beta values from individual subject contrast maps for Near vs Far contrast from the whole-brain GLM fMRI analysis.
Change from baseline in brain activation during non-symbolic number comparison task performance | Baseline and post-intervention (after 6 weeks)
  Neural activity will be measured during functional magnetic resonance imaging (fMRI) non-symbolic number comparison task. Data will consist of beta values from individual subject contrast maps for Near vs Far contrast from the whole-brain general linear model (GLM) fMRI analysis.

SECONDARY OUTCOMES:
Change from baseline in symbolic addition task performance (reaction time) | Baseline and post-intervention (after 6 weeks)
  Performance will be measured by children's reaction time (milliseconds) on symbolic addition task
Change from baseline in symbolic addition task performance (accuracy) | Baseline and post-intervention (after 6 weeks)
  Performance will be measured by children's accuracy (% trials correct) on symbolic addition task

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Cognitive and Systems Neuroscience Laboratory, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No